CLINICAL TRIAL: NCT02646644
Title: Heterogeneity of Metastatic Neuroendocrine Tumors as Determined With 18F-dihydroxyphenylalanine-PET /CT, a Retrospective Analysis
Acronym: HET-NET
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201501247
Record Dates: First submitted 2015-12-24; First posted 2016-01-06 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastasized intestinal NET: We will select the 18F- DOPA-PET scans conducted in the Universtiy Medical Center of Groningen (UMCG) of adult patients with a metastasized intestinal NET between February 2014 until November 2015. Only patients of whose clinical data are available within the UMCG are included.
  Interventions: Other: Metastasized intestinal NET

INTERVENTIONS:
Other: Metastasized intestinal NET — This is an observational study

SUMMARY:
In an individual cancer patient extensive genetic and phenotypic variation exists between and within tumor lesions. Tumour load in NET patients can be measured with fluorine-18-L-dihydroxyphenylalaninepositron emission tomography (18F-DOPA-PET) scan.

This aim of the study is to investigate heterogeneity between tumor lesions within patients with intestinal NET by determining the differences in tracer uptake measured on a 18F- DOPA-PET scan retrospectively.

DETAILED DESCRIPTION:
In an individual cancer patient extensive genetic and phenotypic variation exists between and within tumor lesions. Tumour load in NET patients can be measured with fluorine-18-L-dihydroxyphenylalanine positron emission tomography (18F-DOPA-PET) scan.

This aim of the study is to investigate heterogeneity between tumor lesions within patients with intestinal NET by determining the differences in tracer uptake measured on a 18F- DOPA-PET scan in retrospect.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* diagnosis of intestinal NET diagnosed by a dedicated NET specialist
* more than one positive lesion on the 18F-DOPA-PET scan.
* available CT-scan within 6 months before or after the 18F-DOPA-PET-scan.

Exclusion Criteria:

* no clinical data available at the UMCG, besides the results of the DOPA PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will select the 18F- DOPA-PET scans conducted in the UMCG of adult patients with a metastasized intestinal NET between February 2014 until November 2015. Only patients of whose clinical data are available within the UMCG are included.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
tracer uptake in tumor lesions within patients with intestinal NET | at the day of scan
  The difference in tracer uptake of tumor lesions within patients with intestinal NET measured on a 18F- DOPA-PET scan.

SECONDARY OUTCOMES:
tracer uptake in tumor lesions within patients with intestinal NET adjusted for uptake of background organ | at the day of scan
  The difference in tracer uptake of tumor lesions adjusted for uptake of background organ within patients with intestinal NET measured on a 18F- DOPA-PET scan.

OTHER OUTCOMES:
the correlation of the magnitude of heterogeneity with ki 67 | date of diagnosis until date of scan
  the correlation of the magnitude of heterogeneity between tumor lesions within patients with Intestinal NET, with the ki67 index of the tumor

CONTACTS AND LOCATIONS:
Overall Officials: A. M.E. Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No